CLINICAL TRIAL: NCT00200252
Title: Intramuscular Versus Intravascular Oxytocin for the Third Stage of Labour
Brief Title: Oxytocin Administration in the Third Stage of Labour - A Study of Appropriate Route and Dose
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Memorial University of Newfoundland (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIC05.79
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Third Stage of Labour
Keywords: oxytocin; third stage; dose; route; blood loss
MeSH Terms: conditions — Hemorrhage | interventions — Oxytocin

ARMS (3):
- group B (Active Comparator): women in group B will receive 10 uts oxytocin IM
  Interventions: Drug: oxytocin
- group C (Active Comparator): women in group C will receive oxytocin 5 uts IV
  Interventions: Drug: oxytocin
- group A (Active Comparator): women in group A will receive oxytocin 5 uts IM
  Interventions: Drug: oxytocin

INTERVENTIONS:
Drug: oxytocin

SUMMARY:
Mothers are given the medication oxytocin after birth to help the uterus (womb) contract and therefore reduce blood loss. In Canada, oxytocin is given either into the muscle of the thigh or into a vein. However, it is not known which route is better.This study will test which dose and route of oxytocin is best in reducing blood loss following vaginal delivery.

ELIGIBILITY:
Inclusion Criteria:

* women 19 years and older
* singleton pregnancy
* 32 weeks gestation
* spontaneous vaginal delivery

Exclusion Criteria:

* previous postpartum hemorrhage
* placenta previa
* grand multiparity (>4)
* anticoagulation therapy
* delivery prior to 32 weeks gestation
* operative vaginal delivery
* antepartum hemorrhage > 20 weeks
* hemoglobin <10g/dL
* multiple gestation
* intrauterine death

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2005-09; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
change in hematocrit

SECONDARY OUTCOMES:
estimated blood loss
postpartum hemorrhage (estimated blood loss > 500cc)
severe postpartum hemorrhage (estimated blood loss > 1000cc)
incidence of hypotension
length of third stage of labour
need for blood transfusion
incidence of retained placenta
need for dilatation and curettage
need for hysterectomy
need for additional oxytocics after delivery
postpartum antibiotic use
maternal satisfaction
bleeding needing readmission

CONTACTS AND LOCATIONS:
Overall Officials: Colleen L Cook, MD, Principal Investigator — Resident, Discipline Obstetrics and Gynecology, Memorial University of Newfoundland; Joan Crane, MD, Study Director — Faculty, Discipline Obstetrics and Gynecolgy, Memorial University of Newfoundland
Locations (1):
- Women's Health Centre, Eastern Health, St. John's, Newfoundland and Labrador, Canada

REFERENCES:
- [Derived] Oladapo OT, Okusanya BO, Abalos E, Gallos ID, Papadopoulou A. Intravenous versus intramuscular prophylactic oxytocin for the third stage of labour. Cochrane Database Syst Rev. 2020 Nov 9;11(11):CD009332. doi: 10.1002/14651858.CD009332.pub4. PMID 33169839